CLINICAL TRIAL: NCT05648435
Title: Proximal Tubule Function in Septic Patients as Measured by Endogenous Lithium Clearance
Brief Title: Lithium Clearance in Patients With High Risk of Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: REK 536547
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Urine and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis patients: No interventions
  Interventions: Diagnostic Test: Lithium measures
- Healthy controls: No interventions
  Interventions: Diagnostic Test: Lithium measures

INTERVENTIONS:
Diagnostic Test: Lithium measures — Measurements of lithium levels in blood and urine

SUMMARY:
Renal lithium clearance is hypothesized to be a useful indicator of renal tubular function.

In this study lithium clearance will be monitored in patients with sepsis associated acute kidney injury and in healthy controls.

DETAILED DESCRIPTION:
Lithium is almost completely reabsorbed in the proximal tubule in parallel with sodium and water. What is not reabsorbed here is assumed to be fully excreted in urine, giving a reasonably accurate measurement of sodium reabsorption in the proximal tubule. Endogenous lithium clearance will be measured by inductively coupled plasma mass spectrometry (ICP-MS). The Gomez equations will be applied to calculate efferent arteriolar resistance, afferent arteriolar resistance, glomerular hydrostatic pressure, glomerular filtration pressure, and glomerular oncotic pressure. N-acetyl-β-D glucosaminidase (NAG) and NGAL, markers of tubular injury, will be measured by a spectrophotometric method using a commercially available kit. Routine blood and urine analyses will be performed at the Diagnostic Clinic Laboratory, University Hospital of North Norway, Tromsø.

ELIGIBILITY:
Inclusion criteria sepsis associated acute kidney injury:

* Sepsis diagnosed or suspected
* Age >18 years

Inclusion Criteria healthy controls:

* Previously healthy individuals
* Age >18 years

Exclusion Criteria:

Oliguria or renal impairment due to other causes than sepsis. Pregnancy or breast-feeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intensive care patients and healthy controls
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Renal lithium clearance | Repeated measures between 07:00-20:00
  Measurement of renal lithium clearance at 8AM, 2 PM, and 8 PM

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No